CLINICAL TRIAL: NCT00709696
Title: Human Laboratory Study Of Varenicline in Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 0702M02324; K01DA019446 (NIH); DPMCDA (Other: NIDA)
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Results first posted 2017-12-27 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Nicotine Dependence
Keywords: Tobacco; nicotine; smoking; varenicline; human laboratory study; stress tolerance; startle response; cognitive assessment; progressive ratio
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo Varenicline
  Interventions: Drug: Placebo
- 2 (Active Comparator): Varenicline
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Placebo — Days 1 - 3 (0.5 mg tablet, q.d.), Days 4 - 7 (0.5 mg tablet, b.i.d.), and Day 8 - 21 (1 mg tablet, b.i.d.).
  Other Names: Chantix
  Arms: 1
Drug: Varenicline — Days 1 - 3 (0.5 mg tablet, q.d.), Days 4 - 7 (0.5 mg tablet, b.i.d.), and Day 8 - 21 (1 mg tablet, b.i.d.).
  Other Names: Chantix
  Arms: 2

SUMMARY:
The purpose of this study is to test the ways that a drug called varenicline helps smokers to quit smoking. Varenicline is also called Chantix® and is approved by the United States Food and Drug Administration (FDA) to help people quit smoking. We will test how varenicline works by having you quit smoking and complete tasks that assess how you think and feel. We predict that varenicline help reduce anxiety, improve attention and concentration, and reduce how satisfying cigarettes are.

DETAILED DESCRIPTION:
The purpose of this study is to understand the therapeutic mechanisms of varenicline, a novel nicotinic analogue, through focused measures of potential psychological and physiological mediators. Varenicline is an FDA-approved pharmacotherapy for smoking cessation that is believed to provide relief from craving and withdrawal through agonism and antagonism of some central nervous system nicotinic acetylcholinergic receptors. However, no controlled studies have established the physiological and psychological processes that mediate the efficacy of varenicline in humans. The main goal of the proposed pilot study is to evaluate and compare the effects of varenicline on subjective, cognitive, and physiological outcomes, using a randomized, placebo-controlled, double-blind between-groups design. The study will combine both brief clinical trial methodology with human laboratory approaches. A secondary goal is to validate the utility of the laboratory paradigms for the identification of future smoking cessation agents.

ELIGIBILITY:
Inclusion Criteria:

1.1. Who. Subjects will be women and men between the ages of 18 and 40 who have smoked at least 10 cigarettes per day for at least 1 year. They will respond to requests in the public media for individuals who are interested in quitting smoking.

1.2. Total sample/Number per group. The total randomized sample size will equal 20 subjects, equally distributed across the two medication groups.

1.3. Inclusion Criteria.

1. 18 years to 60 years.
2. Smoke Marlboro Lights (This criterion was selected to reduce inter-subject variation in response variables as has been done in many human laboratory studies of smoking behavior. Over 40% of all smokers smoke some type of the Marlboro brand of cigarette (Substance Abuse and Mental Health Services Administration, 2005). Based on telephone screen data for 767 subjects collected at TURC, Marlboro Light cigarettes are the most common type of Marlboro smoked in our sampling population (158/252 Marlboro users [63%]). Therefore, we have decided to only enroll those smoking Marlboro Light cigarettes, non-menthol).
3. Smoked at least 10 cigarettes/day for at least 1 year.
4. English speaking and reading.
5. Females who are of childbearing potential must practice effective contraception and meet the following criteria:

   1. Are instructed to avoid pregnancy through 30 days after the last dose of study medication.
   2. Have a negative urine pregnancy test at baseline.
   3. Agree to use of the birth control methods listed: an oral contraceptive agent, an intrauterine device (IUD), an implantable contraceptive (e.g., Norplant), or an injectable contraceptive (e.g., Depo-Provera) for at least one month prior to entering the study and will continue its use through at least 30 days after the last dose of the study medication. A barrier method of contraception (e.g., condom or diaphragm with spermicide) while participating in the study and 30 days after the last dose of study medication.
6. Willingness to not use illicit drugs during study period including marijuana.

Exclusion Criteria:

1. Concurrent use of tobacco products (other than cigarettes) or nicotine products.
2. Medications that might affect the outcome measures of nicotine reward, cognition, anxiety, and stress will also be a basis for exclusion. These medications include psychotropic drugs (i.e., anti-psychotic, anti-depressant, anti-anxiety, or stimulant), anti- hypertensive agents (e.g., beta-blockers), and other drugs that can influence the outcome domains.
3. History of kidney disease or renal impairment since varenicline is primarily excreted by the kidney and thus such patients are vulnerable to increased and potentially toxic levels of varenicline.
4. Treatment for drug or alcohol dependence during the last year, or evidence of alcohol abuse so severe that the patient is judged potentially unable to comply with the protocol.
5. Suicidal or homicidal ideation.
6. History of bipolar disorder, schizophrenia, schizoaffective disorder, attention deficit disorder, or attention deficit hyperactivity disorder.
7. Current major depression or anxiety disorder.
8. Pregnant or lactating or planning pregnancy during treatment period.
9. Having plans to leave the immediate geographical area within 2 months.
10. Unwillingness or inability to give written informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2008-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc E Mooney, Ph.D., Principal Investigator — University of Minnesota; Andrew Oliver, B.A., Study Director — University of Minnesota
Locations (1):
- Tobacco Use Research Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Tonstad S, Tonnesen P, Hajek P, Williams KE, Billing CB, Reeves KR; Varenicline Phase 3 Study Group. Effect of maintenance therapy with varenicline on smoking cessation: a randomized controlled trial. JAMA. 2006 Jul 5;296(1):64-71. doi: 10.1001/jama.296.1.64. PMID 16820548
- [Background] Oncken C, Gonzales D, Nides M, Rennard S, Watsky E, Billing CB, Anziano R, Reeves K. Efficacy and safety of the novel selective nicotinic acetylcholine receptor partial agonist, varenicline, for smoking cessation. Arch Intern Med. 2006 Aug 14-28;166(15):1571-7. doi: 10.1001/archinte.166.15.1571. PMID 16908789
- [Background] Nides M, Oncken C, Gonzales D, Rennard S, Watsky EJ, Anziano R, Reeves KR. Smoking cessation with varenicline, a selective alpha4beta2 nicotinic receptor partial agonist: results from a 7-week, randomized, placebo- and bupropion-controlled trial with 1-year follow-up. Arch Intern Med. 2006 Aug 14-28;166(15):1561-8. doi: 10.1001/archinte.166.15.1561. PMID 16908788
- [Background] Jorenby DE, Hays JT, Rigotti NA, Azoulay S, Watsky EJ, Williams KE, Billing CB, Gong J, Reeves KR; Varenicline Phase 3 Study Group. Efficacy of varenicline, an alpha4beta2 nicotinic acetylcholine receptor partial agonist, vs placebo or sustained-release bupropion for smoking cessation: a randomized controlled trial. JAMA. 2006 Jul 5;296(1):56-63. doi: 10.1001/jama.296.1.56. PMID 16820547
- [Background] Gonzales D, Rennard SI, Nides M, Oncken C, Azoulay S, Billing CB, Watsky EJ, Gong J, Williams KE, Reeves KR; Varenicline Phase 3 Study Group. Varenicline, an alpha4beta2 nicotinic acetylcholine receptor partial agonist, vs sustained-release bupropion and placebo for smoking cessation: a randomized controlled trial. JAMA. 2006 Jul 5;296(1):47-55. doi: 10.1001/jama.296.1.47. PMID 16820546
- [Background] Nakamura M, Oshima A, Fujimoto Y, Maruyama N, Ishibashi T, Reeves KR. Efficacy and tolerability of varenicline, an alpha4beta2 nicotinic acetylcholine receptor partial agonist, in a 12-week, randomized, placebo-controlled, dose-response study with 40-week follow-up for smoking cessation in Japanese smokers. Clin Ther. 2007 Jun;29(6):1040-56. doi: 10.1016/j.clinthera.2007.06.012. PMID 17692720
- [Background] Tsai ST, Cho HJ, Cheng HS, Kim CH, Hsueh KC, Billing CB Jr, Williams KE. A randomized, placebo-controlled trial of varenicline, a selective alpha4beta2 nicotinic acetylcholine receptor partial agonist, as a new therapy for smoking cessation in Asian smokers. Clin Ther. 2007 Jun;29(6):1027-39. doi: 10.1016/j.clinthera.2007.06.011. PMID 17692719
- [Background] Williams KE, Reeves KR, Billing CB Jr, Pennington AM, Gong J. A double-blind study evaluating the long-term safety of varenicline for smoking cessation. Curr Med Res Opin. 2007 Apr;23(4):793-801. doi: 10.1185/030079907x182185. PMID 17407636
- [Background] Aubin HJ, Bobak A, Britton JR, Oncken C, Billing CB Jr, Gong J, Williams KE, Reeves KR. Varenicline versus transdermal nicotine patch for smoking cessation: results from a randomised open-label trial. Thorax. 2008 Aug;63(8):717-24. doi: 10.1136/thx.2007.090647. Epub 2008 Feb 8. PMID 18263663
- [Background] Niaura R, Hays JT, Jorenby DE, Leone FT, Pappas JE, Reeves KR, Williams KE, Billing CB Jr. The efficacy and safety of varenicline for smoking cessation using a flexible dosing strategy in adult smokers: a randomized controlled trial. Curr Med Res Opin. 2008 Jul;24(7):1931-41. doi: 10.1185/03007990802177523. Epub 2008 May 29. PMID 18513462
- [Background] Nides M, Glover ED, Reus VI, Christen AG, Make BJ, Billing CB Jr, Williams KE. Varenicline versus bupropion SR or placebo for smoking cessation: a pooled analysis. Am J Health Behav. 2008 Nov-Dec;32(6):664-75. doi: 10.5555/ajhb.2008.32.6.664. PMID 18442345
- [Background] Stapleton JA, Watson L, Spirling LI, Smith R, Milbrandt A, Ratcliffe M, Sutherland G. Varenicline in the routine treatment of tobacco dependence: a pre-post comparison with nicotine replacement therapy and an evaluation in those with mental illness. Addiction. 2008 Jan;103(1):146-54. doi: 10.1111/j.1360-0443.2007.02083.x. Epub 2007 Nov 19. PMID 18028247

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo Varenicline
  Placebo: Days 1 - 3 (0.5 mg tablet, q.d.), Days 4 - 7 (0.5 mg tablet, b.i.d.), and Day 8 - 21 (1 mg tablet, b.i.d.).
- Varenicline: Varenicline
  Varenicline: Days 1 - 3 (0.5 mg tablet, q.d.), Days 4 - 7 (0.5 mg tablet, b.i.d.), and Day 8 - 21 (1 mg tablet, b.i.d.).
Period: Overall Study
Arm/Group | Placebo | Varenicline
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treatment seeking cigarette smokers
Groups:
- Placebo Varenicline: Placebo Varenicline
  Placebo: Days 1 - 3 (0.5 mg tablet, q.d.), Days 4 - 7 (0.5 mg tablet, b.i.d.), and Day 8 - 21 (1 mg tablet, b.i.d.).
- Total: Total of all reporting groups
Arm/Group | Placebo Varenicline | Varenicline | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (5.69) | 38.3 (9.7) | 32.0 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Nicotine Withdrawal Scale
Description: Scale is equal to days subject did not smoke Scale is 0-5 0 being no days 5 being did not quit at all
Time Frame: 21 days
Population: Treatment-seeking smokers
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Varenicline | Varenicline
Number analyzed (Participants) | 4 | 3
units on a scale | 3.3 (5.3) | 0.3 (3.8)

ADVERSE EVENTS:
Arm/Group | Placebo Varenicline | Varenicline
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No